CLINICAL TRIAL: NCT05020522
Title: A Comparison of the Diagnostic Accuracy of Luminal Index Magnetic Resonance Imaging and Multi-parametric Magnetic Resonance Imaging for the Accelerated Detection of Significant Prostate Cancer
Brief Title: Comparison of Diagnostic Accuracy of Luminal Index and MP MRI for Accelerated deTEction of Significant Prostate Cancer
Acronym: CLIMATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 281621
Record Dates: First submitted 2021-07-12; First posted 2021-08-25 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: Magnetic Resonance Imaging; Luminal Index MRI; Methylation Signature; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Paired, non-randomised, comparative study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI scan (Other): Mp-MRI, LI-MRI, plasma DNA methylation signature (optional)
  Interventions: Diagnostic Test: Luminal Index MRI (LI-MRI); Diagnostic Test: LI-MRI targeted prostate biopsy; Diagnostic Test: Plasma methylation signature (ctMethSig)

INTERVENTIONS:
Diagnostic Test: Luminal Index MRI (LI-MRI) — Multiecho T2 sequence; eventual biopsy of lesion(s) detected with LI-MRI only.
Diagnostic Test: LI-MRI targeted prostate biopsy — Biopsy targeted to suspicious lesions detected with LI-MRI only
Diagnostic Test: Plasma methylation signature (ctMethSig) — Blood sample.

SUMMARY:
Multi-parametric (mp) MRI has now internationally been incorporated as standard of care in the work-up of participants with suspected prostate cancer. The standard mpMRI protocol requires 30-45 minutes to be performed and has a sensitivity and specificity of approximately 90% and 50% for the detection of clinically significant prostate cancer. Compared to the non-targeted systematic transrectal ultrasound (TRUS) biopsy approach in men with clinically suspected prostate cancer (e.g.: elevated PSA), performing mpMRI as a triage test allows to detect clinically significant cancer in more men (38% vs 26%) and clinically insignificant cancer in less men (9% vs 22%), while avoiding biopsy in roughly one third of men.

However, there is need for improvement in the prostate diagnostic pathway even after incorporation of mp-MRI, specifically mpMRI can miss significant cancer in around 10% of cases and only 50% of positive scans turn out to harbor significant cancer at biopsy. Moreover, the key functional imaging sequence of mp-MRI (i.e.: DWI) often suffers from image artifacts causing difficulty in scan interpretation.

To address these issues the investigators aim to investigate Luminal Index MRI (LI-MRI), a novel method of MR imaging that requires only up to 10 minutes to be performed and doesn't require the use of contrast media. LI-MRI has shown promising results for the characterization of prostate cancer.

In this study the diagnostic performance of LI-MRI and mpMRI for the detection of prostate cancer will be directly compared.

DETAILED DESCRIPTION:
Luminal Index MRI (LI-MRI). LI-MRI is a novel technique that allows the assessment of luminal water fraction (LWF). The normal prostate consists of a glandular lumen and cellular areas; cancer alters the balance of glandular to cellular spaces, reducing the fraction of glandular lumen. This fraction decreases further as the grade of tumor increases. Using a multiecho T2-weighted sequence, investigators can differentiate between long T2 values of the luminal space and the short T2 values of the stromal/epithelial space. The luminal index of an image pixel can be calculated as a fraction of the area of the luminal space to the sum of cellular-stromal and luminal space. Studies have shown a good correlation between LWF and its histological measurement, with potential to detect prostate cancer and predict tumor grade. From the results of preliminary studies, the optimized LI-MRI sequence has been very good at differentiating clinically significant and non-significant tumors.

PURPOSE. The purpose of the study is to compare the diagnostic performance of LI-MRI (up to 10 minutes scan, no contrast required) and mp-MRI (35-40 min scan, intravenous contrast injection required) for the detection of clinically significant prostate cancer.

DESIGN. This is a prospective, multi-centre, paired, non-randomised, comparative study. Patients with clinically suspected prostate cancer that are scheduled for mpMRI as part of their routine diagnostic workup will be asked to participate to the study. All participants will undergo an additional LI-MRI sequence during the clinical scan session. Mp-MRI and LI-MRI images will be interpreted independently by different radiologists, blinded to the results of the other test. Targeted biopsies will be performed for any suspicious lesion (i.e. MRI score 3-4-5) detected with mpMRI and/or LI-MRI, blinded to the source of the lesion. The diagnostic performance of the two techniques will then be assessed using the results of the targeted biopsy.

An optional translational study will also be performed to investigate the ability of DNA methylation signatures in the plasma to identify men at high risk of metastases from high risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men with clinically suspected prostate cancer and referred for prostate MRI
* Willing and able to provide a written informed consent

Exclusion Criteria:

* Prostate specific antigen (PSA) level > 20ng/ml within 6 months
* Previous diagnosis of prostate cancer
* Ongoing hormone treatment within 3 months prior to MRI, excluding antiandrogens or 5-alpha reductase inhibitors
* Contraindication to MRI scan
* Contraindication to administration of gadolinium-based contrast agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of mp-MRI and LI-MRI | 3 years
  Comparison of per-participant diagnostic accuracy of mp-MRI and LI-MRI for the detection of clinically significant prostate cancer (i.e. Gleason 3+4 or higher). Two endpoints are included in the primary outcome: difference in sensitivity and difference in specificity.

SECONDARY OUTCOMES:
Diagnostic accuracy of LI-MRI as an add-on test | 3 years
  Per-participant diagnostic accuracy of LI-MRI as an add-on test in combination with mp-MRI for the detection of clinically significant cancer.
Proportion of correct clinical recommendation | 3 years
  Comparison of the proportion of men who would receive a correct clinical recommendation that biopsy could be avoided using mp-MRI and LI-MRI by retrospective analysis.
Per-lesion diagnostic accuracy of mp-MRI and LI-MRI | 3 years
  Comparison of per-lesion diagnostic accuracy of LI-MRI and mp-MRI for clinically significant cancer (difference in sensitivity and specificity).
Proportion of non-significant cancer detection | 3 years
  Comparison of the proportion of men diagnosed with non-significant cancer (Gleason 3+3) based on LI-MRI and mp-MRI targeted biopsies.
Value of MRI in diagnostic models | 3 years
  Evaluation of the added value of MRI when included in a diagnostic model of clinically significant cancer based on the clinical features of age and PSA density.
Luminal Index quantitative analysis | 3 years
  Correlation between Luminal Index quantitative metric and tumor Gleason grade
Interobserver agreement on LI-MRI scores | 3 years
  Interobserver agreement among radiologists on LI-MRI scores.
Interobserver agreement on Gleason scores | 3 years
  Interobserver agreement among histopathologists on Gleason scores at biopsy.
ctMethSig true positive rate | 3 years
  Proportion of men with clinically significant cancer who are positive with ctMethSig.
ctMethSig false positive rate | 3 years
  Proportion of men without clinically significant cancer who are positive with ctMethSig.

OTHER OUTCOMES:
ctMethSig and risk of metastases | 3 years
  Correlation of ctMethSig with other clinical factors known to be associated with risk of metastasis (e.g. Gleason grade)

CONTACTS AND LOCATIONS:
Overall Officials: Shonit Punwani, Principal Investigator — University College, London
Locations (1):
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Hammouri T, Brembilla G, Brizmohun M, Tuazon J, Clemente J, Mathew M, Potyka I, Brew-Graves C, Markus J, Giganti F, Parry T, Haider A, Mallett S, Dudderidge T, Barrett T, Attard G, Moore C, Punwani S; CLIMATE Trial Management Group. The 'Comparison of diagnostic accuracy of Luminal Index and standard of care MRI for Accelerated deTEction of prostate cancer' (CLIMATE) trial protocol. BJU Int. 2026 Jan 25. doi: 10.1111/bju.70108. Online ahead of print. PMID 41582606